CLINICAL TRIAL: NCT06665594
Title: Does TXA Reduce Bruising After Hyaluronic Acid Filler Injection? A Prospective Half Face Study
Brief Title: Effect of TXA on Reducing Bruising After Filler Injection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1103; A539730 (Other: UW- Madison); Protocol Version 8/13/25 (Other: UW- Madison)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Facial Filler Injections; Hyaluronic Acid; Tranexamic Acid
MeSH Terms: interventions — Hyaluronic Acid; Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Facial Filler Injection (Experimental): TXA plus HA injection in half of face, saline plus HA injection on other half of face
  Interventions: Procedure: Hyaluronic Acid (HA); Drug: Tranexamic Acid (TXA); Drug: Saline (placebo)

INTERVENTIONS:
Procedure: Hyaluronic Acid (HA) — Injectable gel
Drug: Tranexamic Acid (TXA) — Injection of TXA
Drug: Saline (placebo) — Injection of saline

SUMMARY:
The goal of this clinical trial is to look at the effect tranexamic acid (TXA) may have on reducing bruising, swelling, and pain after facial filler injection. The main question it aims to answer is:

* Does the addition of TXA to hyaluronic acid (HA) reduce bruising, swelling, and tenderness after HA injection?

Participants will receive the study medication along with the standard facial filler injection and complete surveys.

DETAILED DESCRIPTION:
The overall purpose of this study is to evaluate the safety and efficacy of co-administration of TXA with HA in reducing swelling, bruising and pain after facial injection. Researchers will do this by comparing HA to HA+TXA in participants undergoing facial filler injections. Participants undergoing facial filler injections almost always have the same type of injection performed bilaterally in order to maintain symmetry. This provides a unique opportunity where participants can serve as their own controls. Therefore, researchers have designed this as a half face study. Participants will be injected with HA on half of their face and the other half of the face will be injected with HA+TXA. Researchers will then assess swelling, bruising, pain, and overall satisfaction using participant self-reported surveys, physician surveys, and review of medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 but less than or equal to 89 years.
* Participants interested in facial filler (HA) injection.
* English speaking.

Exclusion Criteria:

* Minors or under the age of 18
* Participant over the age of 89
* Pregnant or breast-feeding women
* Individuals unable to give consent due to another condition such as impaired decision-making capacity.
* Individuals with a history of a thrombotic event (DVT, PE, stroke, MI) or genetic disorder that increases risk of thrombosis
* Participants undergoing unilateral facial filler (HA) injection
* Participants with history of hypersensitivity to TXA or any of the other ingredients
* Participants that are on current therapeutic anticoagulation therapy and aspirin use
* Participants with stage 2 or greater renal failure
* Participants on hemodialysis or peritoneal dialysis
* History of diabetes or seizures
* Current tobacco smokers
* Acquired defective color vision

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Intensity of bruising on TXA + HA half of face | Post-procedure day 7
  Participants will score the intensity of bruising on a 5-point Likert scale, where 1 = no bruising and 5 = severe bruising.
Intensity of bruising on saline + HA half of face | Post-procedure day 7
  Participants will score the intensity of bruising on a 5-point Likert scale, where 1 = no bruising and 5 = severe bruising.
Duration of bruising on TXA + HA half of face | Post-procedure day 7
  Participants will indicate on what day their bruising disappeared, or whether it is still there.
Duration of bruising on saline + HA half of face | Post-procedure day 7
  Participants will indicate on what day their bruising disappeared, or whether it is still there.

SECONDARY OUTCOMES:
Intensity of bruising on TXA + HA half of face | Post-procedure day 1
  Participants will score the intensity of bruising on a 5-point Likert scale, where 1= no bruising and 5= severe bruising.
Intensity of bruising on saline + HA half of face | Post-procedure day 1
  Participants will score the intensity of bruising on a 5-point Likert scale, where 1= no bruising and 5= severe bruising.
Duration of bruising on TXA + HA half of face | Post-procedure day 1
  Participants will indicate on what day their bruising disappeared, or whether it is still there.
Duration of bruising on saline + HA half of face | Post-procedure day 1
  Participants will indicate on what day their bruising disappeared, or whether it is still there.
Intensity of swelling on TXA + HA half of face | Post-procedure days 1 and 7
  Participants will score the intensity of swelling on a 5-point Likert scale, where 1 = no swelling and 5 = severe swelling.
Intensity of swelling on saline + HA half of face | Post-procedure days 1 and 7
  Participants will score the intensity of swelling on a 5-point Likert scale, where 1 = no swelling and 5 = severe swelling.
Intensity of pain on TXA + HA half of face | Post-procedure days 1 and 7
  Participants will score the intensity of pain on a 10-point Likert scale, where 0 = no pain and 10 = worst pain possible.
Intensity of pain on saline + HA half of face | Post-procedure days 1 and 7
  Participants will score the intensity of pain on a 10-point Likert scale, where 0 = no pain and 10 = worst pain possible.
Overall satisfaction with aesthetic of TXA + HA half of face | Post-procedure days 1 and 7
  Participants will rate their overall satisfaction on a 5-point Likert scale where 1 = completely dissatisfied and 5 = completely satisfied
Overall satisfaction with aesthetic of saline + HA half of face | Post-procedure days 1 and 7
  Participants will rate their overall satisfaction on a 5-point Likert scale where 1 = completely dissatisfied and 5 = completely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cho, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No